CLINICAL TRIAL: NCT07312500
Title: Application of Fecal DNA Methylation and Fecal Helicobacter Pylori Gastric Cancer Susceptibility Genes in Clinical Diagnosis, Treatment, and Relapse and Metastasis of Gastric Cancer
Brief Title: Fecal DNA Methylation and Helicobacter Pylori SNPs Tests for Gastric Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Director of the gastric surgery department, Fudan University
Other Study IDs: 2410-Exp092-02
Record Dates: First submitted 2025-06-21; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Gastric (Stomach) Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: fecal methylation site-based testing and fecal Helicobacter pylori gastric cancer susceptibility gene-based testing — To establish an early diagnostic test system for gastric cancer based on the methylation site detection technology in feces, with or without the combination of Helicobacter pylori gastric cancer susceptibility gene detection, and then to evaluate the clinical diagnostic value of this test system.

SUMMARY:
Based on the detection technology of methylation sites in feces, combined or not combined with Helicobacter pylori gastric cancer susceptibility gene detection, an early diagnosis and detection system for gastric cancer is established, and the clinical diagnostic value of the detection system is evaluated. In addition, the study observed the association between different loci and post-treatment recurrence, metastasis, or long-term survival rate through long-term follow-up of gastric cancer patients; Follow up with individuals with benign diseases such as gastritis and healthy individuals, compare cases of gastric cancer, and compare their sample data during follow-up with controls who did not have the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female not limited.
2. Within 90 days, the gastroscopy and/or pathological results confirm the absence of gastric cancer.
3. Patients must be able to fully understand the informed consent form and be able to personally sign it.

Exclusion Criteria:

1. Severe heart, liver, kidney dysfunction, or mental illness.
2. History of malignant tumors in the upper gastrointestinal tract.
3. Pregnant women.
4. Those with unclear pathology.
5. Those with unsatisfactory sample retention (such as insufficient sample size).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this clinical study were obtained from inpatients and outpatient follow-up patients attending the sub-center. Subjects will be identified by the investigator based on subject entry criteria and informed of the contents of the informed consent form. Subjects will have their feces collected at the time of clinic visit or at the time of physical examination and will be tested for fecal methylated DNA and H. pylori gastric cancer susceptibility genes.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of early diagnosis of gastric cancer | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China